CLINICAL TRIAL: NCT07009197
Title: Effect of Instrument Assisted Soft Tissue Mobilization on Hand Post Surgical Scars in Primary Flexor Tendons Repair in Zone v
Acronym: IASTM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alzahraa labib abdalaziz, principle investigator : alzahraa labib abdalziz, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005611
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Hand Injuries
Keywords: Instrument Assisted Soft Tissue Mobilization; Primary Flexor Tendons Repair; Hand Post Surgical Scars
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Intervention Model Description: instrumented assisted soft tissue mobilization and tradional therapy
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrument Assisted Soft Tissue Mobilization (Experimental): Twenty-one patients will receive instrument-assisted soft tissue mobilization and traditional therapy three times a week for four weeks.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization; Other: traditional therapy
- traditional therapy (Active Comparator): Twenty-one patients will receive traditional therapy three times a week for four weeks.
  Interventions: Other: traditional therapy

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — the treatment will start by disinfect the instrument between patients to avoid transfer of infections. It is recommended to disinfect the instrument with intermediate-level disinfectants (e.g. isopropyl alcohol), then wash it with soap and water to remove any residuals of the chemical disinfectant off the instrument. If the tools contacts blood, bodily fluids, mucous membranes, or non-intact skin then disinfecting it with high-level disinfectant should be done .IASTM will be done at 30-60 degrees angle for 40-120 seconds+ radiational therapy
  Arms: Instrument Assisted Soft Tissue Mobilization
Other: traditional therapy — the patients will receive traditional therapy in the form of ultrasound, scar massage, and stretching exercises.

SUMMARY:
this study will be conducted to investigate the effect of instrument assisted soft tissue mobilization on hand post surgical scars in primary flexor tendons repair in zone v

DETAILED DESCRIPTION:
The hand plays an important role in independent daily living and in communication with the environment. As the most mobile part of the upper extremity, the hand is actively used in everyday life and professional fields. The flexor tendons of the hand are critical for normal hand function. Injury to these tendons can result in absent finger and wrist flexion, and a subsequent loss of overall hand function. The surgical techniques used to repair these tendons have improved in the past few decades, as have the postoperative rehabilitation protocols. In spite of these advances, flexor tendon repairs continue to be plagued by postoperative scar formation, which limits tendon gliding and prevents a full functional recovery. Many different treatment methods can reduce the trauma and surgical scars. Manual scar treatment is one of these methods. Manual scar therapy to be effective requires applying physiological stimuli adequately to the phase of wound healing. Scar tissue therapy is a treatment for reducing pain and functional limitations, improving pliability, reducing hyper-pigmentation, pruritus, fascial adhesions, to reduce scar thickness and smooth surface area. Instrument assisted soft tissue mobilization (IASTM) is a soft-tissue treatment technique where an instrument is used to provide a mobilizing stimulus to positively affect scar tissue and myofascial adhesion.

ELIGIBILITY:
Inclusion Criteria:

* Both sex will be included in this research
* Hand scar in zone v
* Age varying from 20 to 40
* Hand scar formed post primary flexor tendons repair

Exclusion Criteria:

* Vascular injuries requiring arterial repair
* Soft tissue loss
* Fractures
* Tendon in-juries of other zones
* Preexisting problems such as arthritis limiting joint motion
* unhealed wounds or age of scar under 6 weeks

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-05 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
scar assessment | up to four weeks
  Patient and Observer Scar Assessment Scale (POSAS) will be used to assess scar.It consists of two distinct scales: the OSAS and the PSAS. The PSAS consists of six items: scar-related pain, itchiness, colour, stiffness, thickness and irregularity. Each POSAS item has a 10-point scoring system, with 1 representing normal skin and 10 the worst imaginable scar or sensation; these items are summed to obtain a total score ranging from 6 to 60 for each scale. In addition to the POSAS score, both observer and patient give their own overall opinion on the appearance of the scar using a 10-point scale.

SECONDARY OUTCOMES:
range of motion | up to four weeks
  the range of motion (wrist, metacarpophalangeal, proximal and disatal interphalangeal joint)will be assessed by kinovea software.Kinovea provides a tool to manually draw lines and measure angles to assess ROM as the following:Pause the video at the point where maximum movement occurs (e.g., maximum wrist flexion).Use the angle tool to draw two lines corresponding to the bones of the joint. The software will calculate the angle between the lines, giving you a measure of the ROM.
handgrip strength | up to four weeks
  The hand dynamometer will be used to assess hand grip strength.The subject grips the dynamometer with their maximum force for a few seconds (typically 3 to 5 seconds).Avoid jerky movements or changes in posture during the measurement.